CLINICAL TRIAL: NCT02990429
Title: Comparison Between Forced Air and Intravenous Fluid Warmers in Gynecologic Laparoscopic Surgery
Brief Title: Forced Air and Intravenous Fluid Warmers in Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Warunee Boayam, Faculty of Medicine Siriraj Hospital, Siriraj Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 050/2559(EC2)
Record Dates: First submitted 2016-12-03; First posted 2016-12-13 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2018-08

CONDITIONS: Hypothermia; Anesthesia
Keywords: hypothermia; Shivering; Gynecologic laparoscopic surgery; Warming; General anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Forced Air warmer (bair hugger) (Experimental): .
  In groups: A = 45, receiving intraoperative forced air warming( bair hugger). The forced air was delivered at the high setting of 43ºC
  Interventions: Procedure: Forced Air warmer
- Intravenous Fluid Warmer(ranger warmer) (Experimental): In groups:B =45, having intraoperative intravenous fluid via a fluid warmer patients received intravenous fluid via a fluid warmer after induction anesthesia. The device automatically heated fluid up to 41ºC as set point.
  Interventions: Procedure: Intravenous Fluid Warmer

INTERVENTIONS:
Procedure: Forced Air warmer — * record room temperature
  * record core temperature (tympanic membrane)
  * General anesthesia
  * using forced air warmer (bair hugger)
  * Intravenous fluid at room temperature
  * room temperature and core temperature q15 minutes
  * anesthesia finish, stop bair hugger
  * record core temperature before recovery room
  Arms: Forced Air warmer (bair hugger)
Procedure: Intravenous Fluid Warmer — * record room temperature
  * record core temperature (tympanic membrane)
  * General anesthesia
  * using ranger warmer
  * Intravenous fluid at room temperature
  * room temperature and core temperature q15 minutes
  * anesthesia finish, stop ranger warmer
  * record core temperature before recovery room
  Arms: Intravenous Fluid Warmer(ranger warmer)

SUMMARY:
Perioperative hypothermia is a common problem. It has been defined as a core temperature below 36ºC. The reasons why patient undergoing gynecologic laparoscopic surgery has perioperative hypothermia because the reduced metabolic heat production, redistribution of heat from the core to the periphery and impaired thermoregulation (due to anesthetics), use of cool carbon dioxide gas insufflations and surgical irrigation solution, as well as heat loss due to the cool environment. This perioperative problem has been linked to adverse patient outcomes such as myocardial ischemia as hypothermia increases plasma catecholamine, surgical site infection as hypothermia diminishes wound tissue O2 tension and coagulopathy as hypothermia impairs platelet function.

It claims that perioperative heat loss occurs by radiation (60%), convection (25%) and evaporation (10%). This is caused by the difference between peripheral body and ambient temperature, air circulation around the body and vasodilatation.

In daily practice, most anesthesia personnel warm patient peri-operatively by using force air warmer and intravenous fluid warmer.

This study aimed to compare the difference of core and room temperature in patients undergoing gynecologic laparoscopic surgery by using forced air and intravenous fluid warmer

DETAILED DESCRIPTION:
The study was approved from the Siriraj Institutional Review Board (Si-IRB), COA (Certificate of Analysis): Si201/2016 (18/03/2016), and was written informed consent was obtained from all subjects. The study was conducted at the Department of Siriraj Obstetrics and Gynecology.

A total of 90 patients were enrolled in the study between April 2016 and …..2017. All patients underwent general anesthesia for elective gynecologic laparoscopic surgery. Inclusion criteria were patients aged between 18 and 65, elective case, ASA (American Society of Anesthesiologist) physical status class I-III, BMI 25-30 kg/sq.m., surgical time > 90 minutes. Exclusion criteria were the core temperature less than 36ºC or more than 38ºC. Withdrawal or termination criterion was the change of laparoscopic surgery to exploratory laparotomy.

On the day of surgery, participants signed the informed consent and were randomized equally into two groups: A = 45, receiving intraoperative forced air warming and B =45, having intraoperative intravenous fluid via a fluid warmer All patients underwent general anesthesia after application of standard monitors, anesthesia was induced with fentanyl 1-2 mcg/kg or morphine 0.1-0.2 mg/kg., propofol 1.5-2.5 mg/kg, nimbex 1-1.5 mg/kg or atracurium 0.6 mg/kg. Anesthesia was maintained with sevoflurane ,air,O2, supplemented with fentanyl or morphine.

Core temperatures were measured with an electronic thermometer via tympanic membrane. Intraoperatively, core temperatures and room temperatures were measured at 15 minute intervals until the end of surgery .

Postoperative data were measured at 15 minute intervals at the recovery room. Data consisted of vital sign, core temperature, room temperature, shivering, medication requirements and use of heating devices.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1-3, 18-65 years old, BMI 25-30 kg/sq.m., core temperature 36ºC-38ºC, operation more than 90 minutes

Exclusion Criteria:

* turn operation to exploratory laparotomy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The difference of core and room temperature in patients undergoing gynecologic laparoscopic surgery (by using forced air and intravenous fluid warmer) | 1 Year
  To study the difference between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Warunee Boayam, NS, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj hospital
Locations (1):
- Warunee Boayam, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Allen PB, Salyer SW, Dubick MA, Holcomb JB, Blackbourne LH. Preventing hypothermia: comparison of current devices used by the US Army in an in vitro warmed fluid model. J Trauma. 2010 Jul;69 Suppl 1:S154-61. doi: 10.1097/TA.0b013e3181e45ba5. PMID 20622611
- [Background] Brandt S, Oguz R, Huttner H, Waglechner G, Chiari A, Greif R, Kurz A, Kimberger O. Resistive-polymer versus forced-air warming: comparable efficacy in orthopedic patients. Anesth Analg. 2010 Mar 1;110(3):834-8. doi: 10.1213/ANE.0b013e3181cb3f5f. Epub 2009 Dec 30. PMID 20042442
- [Background] Wagner K, Swanson E, Raymond CJ, Smith CE. Comparison of two convective warming systems during major abdominal and orthopedic surgery. Can J Anaesth. 2008 Jun;55(6):358-63. doi: 10.1007/BF03021491. PMID 18566199
- [Background] Rein EB, Filtvedt M, Walloe L, Raeder JC. Hypothermia during laparotomy can be prevented by locally applied warm water and pulsating negative pressure. Br J Anaesth. 2007 Mar;98(3):331-6. doi: 10.1093/bja/ael369. Epub 2007 Jan 26. PMID 17259258
- [Background] Feroe DD, Augustine SD. Hypothermia in the PACU. Crit Care Nurs Clin North Am. 1991 Mar;3(1):135-44. PMID 2043323
- [Background] Witkowski W, Maj J. [Pathophysiology and management of perioperative hypothermia]. Pol Merkur Lekarski. 2006 Jun;20(120):629-34. Polish. PMID 17007255
- [Background] Turner M, Hodzovic I, Mapleson WW. Simulated clinical evaluation of four fluid warming devices*. Anaesthesia. 2006 Jun;61(6):571-5. doi: 10.1111/j.1365-2044.2006.04589.x. PMID 16704592
- [Background] Bernthal EM. Inadvertent hypothermia prevention: the anaesthetic nurses' role. Br J Nurs. 1999 Jan 14-27;8(1):17-25. doi: 10.12968/bjon.1999.8.1.17. PMID 10085808
- [Background] Bennett J, Ramachandra V, Webster J, Carli F. Prevention of hypothermia during hip surgery: effect of passive compared with active skin surface warming. Br J Anaesth. 1994 Aug;73(2):180-3. doi: 10.1093/bja/73.2.180. PMID 7917732
- [Background] Borms SF, Engelen SL, Himpe DG, Suy MR, Theunissen WJ. Bair hugger forced-air warming maintains normothermia more effectively than thermo-lite insulation. J Clin Anesth. 1994 Jul-Aug;6(4):303-7. doi: 10.1016/0952-8180(94)90077-9. PMID 7946366
- [Background] Giesbrecht GG, Ducharme MB, McGuire JP. Comparison of forced-air patient warming systems for perioperative use. Anesthesiology. 1994 Mar;80(3):671-9. doi: 10.1097/00000542-199403000-00026. PMID 8141463
- [Background] Bieberich MT, Van Duren AP. Thermal control and design considerations for a high-performance fluid warmer. Biomed Instrum Technol. 2003 Mar-Apr;37(2):103-12. doi: 10.2345/0899-8205(2003)37[103:TCADCF]2.0.CO;2. PMID 12677748
- [Background] Patel N, Smith CE, Pinchak AC, Hagen JF. Prospective, randomized comparison of the Flotem Iie and Hotline fluid warmers in anesthetized adults. J Clin Anesth. 1996 Jun;8(4):307-16. doi: 10.1016/0952-8180(96)00040-2. PMID 8695135
- [Background] Presson RG Jr, Bezruczko AP, Hillier SC, McNiece WL. Evaluation of a new fluid warmer effective at low to moderate flow rates. Anesthesiology. 1993 May;78(5):974-80. doi: 10.1097/00000542-199305000-00023. PMID 8489069
- [Background] Faries G, Johnston C, Pruitt KM, Plouff RT. Temperature relationship to distance and flow rate of warmed i.v. fluids. Ann Emerg Med. 1991 Nov;20(11):1198-200. doi: 10.1016/s0196-0644(05)81470-2. PMID 1952305
- [Background] Adriani MB, Moriber N. Preoperative forced-air warming combined with intraoperative warming versus intraoperative warming alone in the prevention of hypothermia during gynecologic surgery. AANA J. 2013 Dec;81(6):446-51. PMID 24597006

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT02990429/Prot_SAP_001.pdf